CLINICAL TRIAL: NCT01583608
Title: ABSORB: Initial Clinical Experience With the Everolimus-eluting Bioresorbable Vascular Scaffold (BVS) System in the Treatment of de Novo Native Coronary Artery Lesions - a Surveillance Registry
Brief Title: ABSORB: Postmarketing Surveillance Registry to Monitor the Everolimus-eluting Bioresorbable Vascular Scaffold in Patients With Coronary Artery Disease
Acronym: ASSURE
Status: Completed | Type: Observational
Sponsor: Medical Care Center Prof. Mathey, Prof. Schofer, Ltd. (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Detlef Mathey, Professor Dr. med. D. Mathey, Medical Care Center Prof. Mathey, Prof. Schofer, Ltd.
Other Study IDs: BVS 12
Record Dates: First submitted 2012-04-17; First posted 2012-04-24 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Coronary Restenosis; Heart Diseases; Coronary Stenosis; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: Drug eluting stent; Bioabsorbable; Bioresorbable; Coronary Stent; Scaffold; Stents; Angioplasty; Coronary Artery Disease; Stentthrombosis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Coronary Restenosis; Heart Diseases; Coronary Stenosis; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The registry aims to evaluate the safety, performance and efficacy of the Everolimus-eluting bioresorbable vascular scaffold (BVS) system in patients with de novo native coronary artery lesions in all-day clinical practice.

DETAILED DESCRIPTION:
Bioresorbable scaffolds are transient implants. They act like drug-eluting metallic stents (DES) during the first 3 months by supporting the vessel wall thereby keeping the artery patent. Subsequently, resorption of the scaffold begins and its structure loosens. As a result of everolimus release, neointimal growth is inhibited similar to DES. Finally the implant is reabsorbed completely in about 2-3 years. BVS in terms of late stent thrombosis may be safer than DES. Transiently scaffolded vessels may regain their natural curvature and angulation as well as response to nitroglycerine and endothelial function.

ELIGIBILITY:
The recommendation to implant BVS in an individual patient is purely based on clinical grounds. These are determined by the instructions for use (IFU) of the BVS and by the clinical experience accumulated so far from clinical studies.These studies suggest that the BVS should be implanted under certain conditions, which are determined by the patient and the coronary lesion treated:

Eligible:

Regarding to patient

* Patient ≥ 18 and ≤ 75 years with a live expectancy of at least 5 years with ischemic heart disease (chronic, NSTEMI and unstable angina) due to one or more de novo native coronary artery lesions
* Patients with evidence of myocardial ischemia

Regarding to lesion

* Reference vessel diameter ≥ 2.0 mm and ≤ 3.8 mm, visually estimated and by online QCA
* Percent diameter stenosis ≥ 50% and < 100%, visually estimated and by online QCA
* TIMI ≥1
* Previous interventions of target vessel lesions should have been done ≥ 6 months prior to index procedure and > 10 mm distal to the target lesion
* Previous interventions of non-target vessel lesions should have been done ≥ 30 days prior to index procedure
* In case of >1 target lesions, those should be from different epicardial vessels

Not eligible:

Regarding to patient

* Patient in whom antiplatelet therapy and/or anticoagulant therapy is contraindicated
* Patient with a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, ticlopidine, prasugrel and ticagrelor, everolimus, poly (L-lactide), poly (D,L-lactide), or platinum, or with contrast sensitivity, who cannot be adequately premedicated
* Patient has a known diagnosis of acute myocardial infarction (STEMI) within 72 hours preceding the index procedure and CK and CK-MB have not returned within normal limits at the time of procedure
* Patient is currently experiencing clinical symptoms consistent with STEMI
* Patient has current unstable arrhythmias
* Patient has a known left ventricular ejection fraction < 30%
* Patient has received a heart transplant or any other organ transplant or is waiting for any organ transplant
* Patient receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease
* Patient is receiving or scheduled to receive chronic anticoagulation therapy
* Elective surgery is planned within the first 6 month after the procedure that will require discontinuing either aspirin or clopidogrel
* Patient has a platelet count < 100 000 cells/mm3 or > 700 000 cells/mm3, a WBC of
* < 3000 cells/mm3, or documented or suspected liver disease
* Patient has known renal insufficiency
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has cerebrovascular accident or transient ischemic neurological attack within the past six month
* Patient has had a significant GI or urinary bleed within the past six months
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non.compliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., les than one year)
* Women of childbearing potential who have not undergone surgical sterilization or are not post-menopausal

Regarding to lesion

* Aorto-ostial location
* Left main location
* Located within 2 mm of the origin of LAD or LCX
* Located within an arterial or saphenous vein graft or distal to a diseased (defined as vessel irregularity per angiogram and > 20% stenosed lesion by visual estimation) arterial or saphenous vein graft
* Lesion involving a bifurcation with side branch vessel ≥ 2 mm in diameter, ostial lesion > 40% stenosed by visual estimation or side branch requiring predilation
* Total occlusion (TIMI flow 0), prior to wire passing
* Excessive tortuosity proximal to or within the lesion (extreme angulation (≥ 90°) proximal to or within the lesion)
* Heavy calcification
* Restenotic from previous intervention
* Target vessel is containing thrombus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular disease
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
(This trial has no primary outcome, all outcomes are of equal weight), Major Adverse Cardiac Event (MACE) | at 24 months
  Composite of ischemia driven target lesion revascularisation (TLR), myocardial infarction and cardiac death

SECONDARY OUTCOMES:
Acute procedural success | At the end of hospital stay (maximum of 7 days)
  Achievement of final in-scaffold residual stenosis of < 50% and TIMI flow 3 of the target site. Successful delivery and deployment of at least one study scaffold at the intended target lesion and successful withdrawal of the delivery system for all target lesions without occurrence of cardiac death, target vessel MI or repeat TLR during hospital stay (maximum of 7 days). In dual target lesion setting both lesions must meet clinical procedure success criteria.
Acute device success | At time of intervention
  Successful delivery and deployment of the first scaffold at the intended target lesion (in overlapping setting both planned scaffolds) and successful withdrawal of delivery system. Attainment of < 50 % residual stenosis and TIMI flow 3 of the target site, using the BVS without the need for other non- study stents.
Scaffold thrombosis | At time of intervention, and at 6, 12, 24, 36 months
Cardiac death | At time of intervention, and at 6, 12,24, 36 months
Myocardial infarction | At time of intervention, and at 6, 12, 24 36 months
Ischemia driven target lesion revascularisation (TLR) | At time of intervention, and at 6, 12, 24, 36 months
  Target lesion denominates scaffolded segment and 5 mm beyond.
Major Adverse Cardiac Event (MACE) | At time of intervention, participants will be followed for the duration of hospital stay (an expected average of 3 days), at 6, 12, 36 months
  Composite of ischemia driven target lesion revascularisation (TLR), myocardial infarction and cardial death
Ischemia driven target vessel revascularisation (TVR) | at 6, 12, 24, 36 months
  TVR is ischemia driven.
Ischemia driven target vessel failure (TVF) | at 6, 12, 24, 36 month
In-lesion % diameter stenosis | Prior procedure
In-scaffold % diameter stenosis | At time of intervention and at angiographic FU if applicable
Minimal lumen diameter (MLD) | Prior and post procedure and at FU if applicable
In-scaffold late lumen loss (LLL) | At angiographic follow-up if applicable
Proximal and distal late lumen loss (LLL) | At angiographic follow-up if applicable
In-lesion late lumen loss | At angiographic follow-up if applicable
Response to nitroglycerin | Before scaffold implantation, during angiographic follow-up if applicable
In-lesion angiographic binary restenosis (≥ 50%) | At angiographic follow-up if applicable
Curvature (cm-1) | Prior and post procedure and at angiographic follow-up if applicable
  treated region
Angulation (°) | Prior and post procedure and at angiographic follow-up if applicable
  Treated region
Clinical success | At time of intervention, and at 6, 12, 24, 36 months
  Procedural success and freedom from TVF, TVR, CABG and scaffold thrombosis
Coronary artery bypass grafting (CABG) | at 6, 12, 24, 36 month

CONTACTS AND LOCATIONS:
Overall Officials: Detlef G Mathey, MD, Principal Investigator — Medical Care Center Prof. Mathey, Prof. Schofer GmbH
Locations (6):
- Germany (6):
  - Medical Care Center Prof. Mathey, Prof. Schofer GmbH, Hamburg, Hamburg
  - Herzzentrum Brandenburg in Bernau, Bernau
  - Klinikum Coburg GmbH, Coburg
  - Elisabeth-Krankenhaus Essen GmbH, Essen
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Background] Serruys PW, Onuma Y, Dudek D, Smits PC, Koolen J, Chevalier B, de Bruyne B, Thuesen L, McClean D, van Geuns RJ, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Sudhir K, Garcia-Garcia HM, Ormiston JA. Evaluation of the second generation of a bioresorbable everolimus-eluting vascular scaffold for the treatment of de novo coronary artery stenosis: 12-month clinical and imaging outcomes. J Am Coll Cardiol. 2011 Oct 4;58(15):1578-88. doi: 10.1016/j.jacc.2011.05.050. PMID 21958884
- [Background] Dudek D, Onuma Y, Ormiston JA, Thuesen L, Miquel-Hebert K, Serruys PW. Four-year clinical follow-up of the ABSORB everolimus-eluting bioresorbable vascular scaffold in patients with de novo coronary artery disease: the ABSORB trial. EuroIntervention. 2012 Jan;7(9):1060-1. doi: 10.4244/EIJV7I9A168. PMID 21959320
- [Background] Diletti R, Onuma Y, Farooq V, Gomez-Lara J, Brugaletta S, van Geuns RJ, Regar E, de Bruyne B, Dudek D, Thuesen L, Chevalier B, McClean D, Windecker S, Whitbourn R, Smits P, Koolen J, Meredith I, Li D, Veldhof S, Rapoza R, Garcia-Garcia HM, Ormiston JA, Serruys PW. 6-month clinical outcomes following implantation of the bioresorbable everolimus-eluting vascular scaffold in vessels smaller or larger than 2.5 mm. J Am Coll Cardiol. 2011 Jul 12;58(3):258-64. doi: 10.1016/j.jacc.2011.02.052. PMID 21737016
- [Background] Gomez-Lara J, Brugaletta S, Farooq V, van Geuns RJ, De Bruyne B, Windecker S, McClean D, Thuesen L, Dudek D, Koolen J, Whitbourn R, Smits PC, Chevalier B, Morel MA, Dorange C, Veldhof S, Rapoza R, Garcia-Garcia HM, Ormiston JA, Serruys PW. Angiographic geometric changes of the lumen arterial wall after bioresorbable vascular scaffolds and metallic platform stents at 1-year follow-up. JACC Cardiovasc Interv. 2011 Jul;4(7):789-99. doi: 10.1016/j.jcin.2011.04.009. PMID 21777888